CLINICAL TRIAL: NCT00177593
Title: The Effect of HealthWear on Short-Term Weight Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0503021
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2005-09

CONDITIONS: Weight Loss; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

INTERVENTIONS:
Behavioral: behavioral weight loss

SUMMARY:
The purpose of this study is to examine the effect of a computer tracking system and energy expenditure device on weight loss in adults.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years of age.
2. Body mass index (BMI) between 25.0-39.9 kg/m2.
3. Access to a computer, Internet access, and will demonstrate proficiency with using the Internet and Web-based software programs. Potential participants will be asked to provide the type of computer they have, the name of their internet service provider, and will have to demonstrate their ability to search the internet during their screening visit.

Exclusion Criteria:

1. Report losing >5% of current body weight in the previous 6 months.
2. Report participating in a research project involving weight loss or physical activity in the previous 6 months.
3. For women, report being pregnant during the previous 6 months, or planning on becoming pregnant over the following 3 months of the intervention. (Pregnancy during initial screening will be based on self-report and will be included on the detailed medical history that is completed by subjects. In addition, this will also be obtained as part of the signed medical clearance from the individual's personal physician.)
4. Currently being treated for any medical condition that could impact body weight (i.e., diabetes mellitus, cancer, etc.).
5. History of myocardial infarction, or a history of undergoing heart surgery such as bypass or angioplasty.
6. Taking medication that would affect heart rate or blood pressure responses to exercise (e.g., beta blockers).
7. Taking medication that could affect metabolism and/or contribute to a change in body weight (e.g., synthroid).
8. Being treated by a therapist for psychological issues or problems, taking pyschotropic medications, or receiving treatment with psychotropic medications within the previous 6 months.
9. No exclusion criteria shall be based on race, ethnicity, or gender.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75
Dates: Start 2005-06; Study Completion 2005-09

PRIMARY OUTCOMES:
weight loss

SECONDARY OUTCOMES:
fitness
physical activity
dietary intake
mediators

CONTACTS AND LOCATIONS:
Overall Officials: John M Jakicic, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States